CLINICAL TRIAL: NCT07127536
Title: Effects of the Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach on Occupational Performance and Executive Function in Adults With Stroke: A Randomised Controlled Trial
Brief Title: Effects of the CO-OP Approach on Occupational Performance and Executive Function in Adults With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Damla Aygün Gürbüz, Principal Investigator - PhD Student in Occupational Therapy, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2023-218
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive standard occupational therapy plus the CO-OP (Cognitive Orientation to daily Occupational Performance) approach. CO-OP sessions will be delivered 5 days per week for 4 weeks, with each session lasting 45 minutes. The intervention focuses on improving performance in meaningful daily activities and enhancing cognitive skills.
  Interventions: Behavioral: CO-OP (Cognitive Orientation to daily Occupational Performance)
- Control Group (Active Comparator): Participants in this group will receive standard occupational therapy only, without the additional CO-OP intervention. Therapy sessions will follow the usual care protocols for stroke rehabilitation at the study site.
  Interventions: Behavioral: Standard Occupational Therapy

INTERVENTIONS:
Behavioral: CO-OP (Cognitive Orientation to daily Occupational Performance) — The CO-OP approach is a client-centered, performance-based intervention that uses cognitive strategies to help individuals improve performance in meaningful daily activities. In this study, CO-OP sessions will be delivered in addition to standard occupational therapy, 5 days per week for 4 weeks, with each session lasting 45 minutes. The intervention group will receive standard occupational therapy intervention in addition to CO-OP.
  Standard Occupational Therapy Therapy sessions will follow the usual care protocols for stroke rehabilitation at the study site.
  Arms: Intervention Group
Behavioral: Standard Occupational Therapy — Participants in this group will receive standard occupational therapy only, without the additional CO-OP intervention. Therapy sessions will follow the usual care protocols for stroke rehabilitation at the study site.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to use the Cognitive Orientation to Daily Occupational Performance (CO-OP) approach with people who have experienced a stroke. This method helps individuals improve how they perform daily tasks by teaching them problem-solving strategies.

This study will answer the following main questions:

Does the CO-OP approach help participants perform their daily activities more easily? Does the CO-OP approach support thinking skills such as planning and attention?

Researchers will look at changes in participants' daily activity performance and thinking skills before and after the CO-OP sessions.

Participants will be randomly assigned to one of two groups:

Complete simple tests before and after the sessions Practice real-life daily activities that are meaningful to them Intervention group: Will receive standard occupational therapy plus CO-OP sessions. The CO-OP sessions will take place 5 days a week for 4 weeks, with each session lasting 45 minutes.

Control group: Will receive only standard occupational therapy as part of usual care.

ELIGIBILITY:
Inclusion Criteria:

* Being in the subacute phase after stroke (3 months < stroke onset < 2 years)
* First-ever stroke
* Brunnstrom stage 2 or above
* Ability to read and write
* Receiving rehabilitation services at Ankara Etlik City Hospital, Physical Medicine and Rehabilitation Hospital

Exclusion Criteria:

* Having any orthopedic, psychological, or neurological disorder other than stroke
* Having moderate to severe aphasia
* Having cognitive impairment (Mini-Mental State Examination score ≤ 24)
* Not willing to participate in the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline and 4 weeks after the start of intervention.
  It is an assessment tool used to evaluate individuals' activity performance and satisfaction levels, and to identify problems encountered in daily life through a semi-structured interview. In this assessment, the individual rates their occupations in terms of performance and importance. In the first stage, problems are identified; in the next stage, the individual is asked to rate the importance of the identified occupations on a scale from 1 to 10. In the final stage, the individual selects the five most important activities and rates both performance and satisfaction for these activities on a scale from 1 to 10. Higher scores indicate higher activity performance and satisfaction.

SECONDARY OUTCOMES:
Performance Quality Rating Scale | Baseline and 4 weeks.
  It is a performance-based observational rating scale used to evaluate the actual performance of activities selected by the individual. It is used together with the Canadian Occupational Performance Measure (COPM) to assess the quality of activity performance. The scale is scored from 1 to 10, where a score of 1 indicates that the individual is unable to perform the activity, and a score of 10 indicates that the activity is completed successfully. The activities identified in the COPM are performed without any verbal or physical guidance.
Executive Function Performance Test | Baseline and 4 weeks.
  It is an assessment tool that evaluates the individual's need for assistance while performing simple daily tasks. It examines the execution of four essential instrumental activities of daily living required for self-care and independent living: simple cooking, telephone use, medication management, and bill payment. The test assesses the ability to meet executive function components in all four tasks: (1) task initiation, (2) task execution, and (3) task completion. The level of cueing required to support task performance is recorded on a five-point scale: 0 = no cueing needed, 1 = verbal guidance, 2 = gestural or physical cueing, 3 = direct verbal assistance, 4 = physical assistance, 5 = the examiner performs the task. The scoring range is 0-25 for each task, with a total score ranging from 0 to 100 across all four tasks. Higher scores indicate greater difficulty in executive functioning.
Stroke Impact Scale version-3.0 | Baseline and 4 weeks.
  This scale is designed to evaluate the quality of life after stroke as perceived by patients themselves or their caregivers. It consists of 8 subscales and 59 items. Each item is scored using a 5-point Likert scale based on the level of difficulty experienced during the past week. Scores for each domain range from 0 to 100. In addition, the scale includes a single-item visual analog scale from 0 to 100 to assess perceived recovery after stroke (0 = no recovery, 100 = full recovery). Higher scores indicate better function and less impact of stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP